CLINICAL TRIAL: NCT02244554
Title: Prospective, Open-Label Comparison Study of Picosecond and Nanosecond Pulse Durations Using a Q-switched Nd:YAG Laser for Tattoo Removal
Brief Title: Comparison Study of Picosecond and Nanosecond Pulse Durations Using a Q-switched Nd:YAG Laser for Tattoo Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-14-TPS05
Record Dates: First submitted 2014-07-24; First posted 2014-09-19 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Tattoo Removal
Keywords: tattoo removal; Q-switched laser; Nd:YAG laser; nanosecond laser; picosecond laser; laser therapy; tattoo; pulsed-laser; laser treatment; remove tattoo; tattoo clearing; tattoo lightening; tattoo lighten; resistant tattoo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- enLighten Laser Picosecond Pulse (Experimental): Picosecond Pulse-duration with enLighten Q-switched Nd:YAG (1064 nm and 532 nm) laser treatment
  Interventions: Device: enLighten Laser
- enLighten Laser Nanosecond Pulse (Experimental): Nanosecond Pulse-duration with enLighten Q-switched Nd:YAG (1064 nm and 532 nm) laser treatment
  Interventions: Device: enLighten Laser

INTERVENTIONS:
Device: enLighten Laser — Picosecond pulse-duration or Nanosecond pulse-duration tattoo treatment with enLighten Q-switched Laser Treatment

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of laser tattoo removal with picosecond pulse durations as compared to treatment with nanosecond pulse durations using a single novel Q-Switched (QS) Nd:YAG laser.

DETAILED DESCRIPTION:
This is a randomized, split-tattoo, open-label, single-center study of up to 25 subjects with tattoos containing black or dark blue ink, alone or in combination with other colors. It will compare the safety and efficacy of nanosecond and picosecond pulse durations with the Cutera Picosecond Q-Switched Nd:YAG laser for tattoo removal.

ELIGIBILITY:
Inclusion Criteria:

* Females or Males, 18 to 55 years of age (inclusive).
* Fitzpatrick Skin Type I - VI.
* Tattoos containing black/blue ink alone or in combination with other colors. No tribal, scarred, high-ink density, or highly colorful tattoos.
* Target tattoos older than 1 year.
* Must be able to read, understand and sign the Informed Consent Form.
* Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
* Wiling to cover tattoos with a bandage or clothing; and/or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treated area starting 2 to 4 weeks before the treatment and/or every day for the duration of the study, including the follow-up period.
* Willing to use hydroquinone approximately 4 weeks pre-treatment and post-treatment if required by Investigator.
* Willingness to have digital photographs taken of the treated area.
* Agree not to undergo any other procedure(s) for the tattoo removal during the study.
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study.

Exclusion Criteria:

* Participation in a study of another device or drug within 6 months prior to enrollment or during the study.
* History of allergic reaction to pigments following tattooing.
* Presence of double tattoo in the treatment area or presence of tribal, scarred, high-ink density, or highly colorful single tattoos.
* History of allergy to local anesthetics.
* History of allergy to topical antibiotics.
* History of malignant tumors in the target area.
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles.
* Pregnant and/or breastfeeding.
* Having an infection, dermatitis or a rash in the treatment area.
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
* Suffering from coagulation disorders or taking prescription anticoagulation medications.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* History of vitiligo, eczema, or psoriasis.
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* History of seizure disorders due to light.
* Any use of medication that is known to increase sensitivity to light according to the Investigator's discretion.
* History of herpes simplex and/or herpes zoster (shingles).
* History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Systemic use of corticosteroid within 12 months of study participation.
* Use of oral isotretinoin within 12 months of study participation and topical use of isotretinoin within 6 months on the treated area.
* Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Current smoker or history of smoking within 6 months of study participation.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Victor Ross, MD, Principal Investigator — Scripps Clinic Carmel Valley
Locations (1):
- Scripps Clinic Carmel Valley, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Sides of tattoos treated
Groups:
- All Study Participants: Subject tattoos were divided into 2 sides for assignment into 2 arms for treatment by the Picosecond and Nanosecond Pulse-duration with enLighten Q-switched Nd:YAG (1064 nm and 532 nm) : active control arm and treatment arm. One side will receive treatment with the picosecond pulse duration and one side will receive treatment with the nanosecond pulse duration.
Period: Overall Study
Arm/Group | All Study Participants
Started | 10; 20 Sides of tattoos treated
Treatment With Picosecond Pulse Duration | 10; 10 Sides of tattoos treated
Treatment With Nanosecond Pulse Duration | 10; 10 Sides of tattoos treated
Completed | 10; 20 Sides of tattoos treated
Not Completed | 0; 0 Sides of tattoos treated

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Subjects All Enrolled Subjects: Picosecond and Nanosecond Pulse-duration with enLighten Q-switched Nd:YAG (1064 nm and 532 nm) laser treatment
Arm/Group | All Enrolled Subjects All Enrolled Subjects
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Level of Tattoo Clearing at 12 Weeks for Each Treatment Arm as Assessed by the Blinded Reviewers.
Description: Physician's Global Assessment (min=0; Max=4) Higher scores indicate better outcomes
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- enLighten Laser Picosecond Pulse: Picosecond Pulse-duration with enLighten Q-switched Nd:YAG (1064 nm and 532 nm) laser treatment
  enLighten Laser: Picosecond pulse-duration pulse-duration tattoo treatment with enLighten Q-switched Laser Treatment
- enLighten Laser Nanosecond Pulse: Nanosecond Pulse-duration with enLighten Q-switched Nd:YAG (1064 nm and 532 nm) laser treatment
  enLighten Laser: Nanosecond pulse-duration tattoo treatment with enLighten Q-switched Laser Treatment
Arm/Group | enLighten Laser Picosecond Pulse | enLighten Laser Nanosecond Pulse
Number analyzed (Participants) | 10 | 10
score on a scale | 3 (.94) | 3 (.82)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | enLighten Laser Picosecond Pulse | enLighten Laser Nanosecond Pulse
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | enLighten Laser Picosecond Pulse (N=10) | enLighten Laser Nanosecond Pulse (N=10)
Erythema (Skin and subcutaneous tissue disorders) | 10 (10) | 10 (10)
Edema (Skin and subcutaneous tissue disorders) | 10 | 10
Purpura (Skin and subcutaneous tissue disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No